CLINICAL TRIAL: NCT02252393
Title: Prospective Randomized Comparison of Intracorporeal Versus Extracorporeal Urinary Diversion During Robotic Radical Cystectomy
Brief Title: Urinary Diversion During Robotic Assisted Radical Cystectomy in Patients With Bladder Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: waiting on surgeon training
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE7814; NCI-2014-01530 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CASE 7814 (Other: Case Comprehensive Cancer Center); P30CA043703 (NIH)
Record Dates: First submitted 2014-09-26; First posted 2014-09-30 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Recurrent Bladder Cancer; Stage 0 Bladder Cancer; Stage I Bladder Cancer; Stage II Bladder Cancer; Urinary Complications
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (RARC with IUD) (Experimental): Patients undergo RARC with IUD.
  Interventions: Procedure: robot-assisted laparoscopic surgery; Other: intraoperative complication management/prevention; Other: quality-of-life assessment
- Arm II (RARC with EUD) (Experimental): Patients undergo RARC with EUD.
  Interventions: Procedure: robot-assisted laparoscopic surgery; Other: intraoperative complication management/prevention; Other: quality-of-life assessment

INTERVENTIONS:
Procedure: robot-assisted laparoscopic surgery — Undergo RARC with IUD
  Arms: Arm I (RARC with IUD)
Procedure: robot-assisted laparoscopic surgery — Undergo RARC with EUD
  Arms: Arm II (RARC with EUD)
Other: intraoperative complication management/prevention — Undergo RARC with IUD
  Arms: Arm I (RARC with IUD)
Other: intraoperative complication management/prevention — Undergo RARC with EUD
  Arms: Arm II (RARC with EUD)
Other: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This randomized clinical trial studies intracorporeal or extracorporeal urinary diversion during robotic assisted radical cystectomy in reducing complications in patients with bladder cancer. Radical cystectomy is surgery to remove the entire bladder as well as nearby tissues and organs. After the bladder is removed, urinary diversion (a surgical procedure to make a new way for urine to leave the body) is performed. It is not yet known whether intracorporeal (within the body) or extracorporeal (outside of the body) urinary diversion is a better method in patients with bladder cancer undergoing robotic assisted radical cystectomy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare perioperative outcomes and complications after robotic assisted radical cystectomy (RARC) with intracorporeal urinary diversion (IUD) and RARC with extracorporeal urinary diversion (EUD) in a prospective randomized fashion.

SECONDARY OBJECTIVES:

I. Time to passage of flatus. II. Analgesic requirement (narcotic use). III. Hospital length of stay. IV. Total operating time. V. Estimated blood loss. VI. Readmission rate. VII. Bladder Cancer Index Questionnaire. VIII. Ureteral strictures. IX. Stomal stenosis. X. Disease recurrence. XI. Secondary procedures.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients undergo RARC with IUD.

ARM II: Patients undergo RARC with EUD.

After completion of study treatment, patients are followed up within 90 days and then for 2-5 years.

ELIGIBILITY:
Inclusion Criteria:

* Grade G1 - G3 bladder cancer
* T stage: cTis - T2
* N0
* M0
* American Society of Anesthesiologists (ASA) < 4
* Informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status 2 or better
* Hemoglobin (Hgb) > 8.0 g/dL
* White blood cell (WBC) > 2.0 k/uL
* Platelets > 50,000
* Creatinine < 3.0 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) < 5.0 x ULN
* Alanine transaminase (ALT) < 5.0 x ULN

Exclusion Criteria:

* Patient unsuitable for or refusing radical cystectomy
* T stage ≥ T3 (mass extending outside the bladder)
* Gross nodal or metastatic disease at presentation (≥ N1, M1)
* Prior pelvic radiation
* Prior open or laparoscopic/robotic bladder or prostate surgery
* Prior colorectal surgery or history of inflammatory bowel disease
* Body mass index (BMI) ≥ 40
* ECOG performance status 3 or worse
* History of coagulopathy or bleeding disorders
* Chronic steroid use
* Patients with end stage renal disease (ESRD) and/or on dialysis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Complication rate | 90 days after surgery
  Analyzed using multivariable logistical regression. Descriptions and grading scales found in the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for adverse event reporting.

SECONDARY OUTCOMES:
Time to passage of flatus | Up to 90 days
  Analyzed using regression analysis.
Analgesic requirement (narcotic use) | Up to 90 days
  Analyzed using logistical regression.
Hospital length of stay | Up to 90 days
  Analyzed using regression analysis.
Total operating time | Up to completion of surgery
  Analyzed using regression analysis.
Estimated blood loss | Up to 90 days
  Analyzed using regression analysis.
Readmission rate | Up to 90 days
  Analyzed using regression analysis.
Quality of life assessed using the Bladder Cancer Index Questionnaire | Up to 5 years
  The Cox proportional hazards model will be used. The hazard ratio (HR) and 95% confidence interval (95% CI) associated with the use of RARC with IUD compared with the use of RARC with EUD will be calculated.
Ureteral strictures | Up to 5 years
  The Cox proportional hazards model will be used. The HR and 95% CI associated with the use of RARC with IUD compared with the use of RARC with EUD will be calculated.
Stromal stenosis | Up to 5 years
  The Cox proportional hazards model will be used. The HR and 95% CI associated with the use of RARC with IUD compared with the use of RARC with EUD will be calculated.
Disease recurrence | Up to 5 years
  The Cox proportional hazards model will be used. The HR and 95% CI associated with the use of RARC with IUD compared with the use of RARC with EUD will be calculated.
Secondary procedures | Up to 5 years
  The Cox proportional hazards model will be used. The HR and 95% CI associated with the use of RARC with IUD compared with the use of RARC with EUD will be calculated.
Cumulative complication incidence | Up to 5 years
  Graphically described using the Kaplan-Meier method. Descriptions and grading scales found in the NCI CTCAE version 4.0 will be utilized for adverse event reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Jihad Kaouk, Principal Investigator — Case Comprehensive Cancer Center